CLINICAL TRIAL: NCT06971822
Title: Assessing the Impact of a Leucine Enriched Whey Protein vs Isonitrogenous Whey on Muscle Protein Synthetic Responses in the Rested and Acute Post Exercise States in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Philip Atherton, Professor Philip Atherton, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AFI3- FMHS 63-0125
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-03

CONDITIONS: Healthy Male Volunteers Over 65
Keywords: Leucine; Muscle Mass; Sarcopenia; Nutrition; Protein
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isonitrogenous Whey Protein Group (Active Comparator): This group will receive a 20g supplement of isonitrogenous whey protein supplement with each of their controlled meals on the study visits.
  Interventions: Dietary Supplement: Protein Supplementation
- BLG (Experimental): This group will receive a 20g supplement of BLG (leucine enriched protein) supplement with each of their controlled meals on the study visits.
  Interventions: Dietary Supplement: Protein Supplementation

INTERVENTIONS:
Dietary Supplement: Protein Supplementation — We are assessing the supplementation of a controlled diet with beta-lactoglobulin protein compared to regular isonitrogenous whey protein. We will make these comparisons over both the 24 hour rested and 24 hour post-exercise states. Beta-lactoglobulin has a higher leucine content than traditional whey protein, with this leucine amino acid thought to have a critical role as an anabolic stimulus to initiate muscle protein synthesis.

SUMMARY:
Occupying ~45-55% of body mass, skeletal muscle is the largest organ of the body and plays a pivotal role in locomotion, structural support and whole-body metabolic health. Additionally, skeletal muscle serves as the largest reservoir of amino acids (AA), which negatively adapts in states of disease and fasting to provide energy and AAs for vital organs, but also positively adapts to nutrition (i.e. protein consumption) and exercise (i.e. resistance exercise (RE)). With the current global ageing population, pressure on health and social care systems is continuing to mount due to increased frailty and other age-related co-morbidities. Sarcopenia, the loss of muscle mass (atrophy) and function with advancing age, predisposes an individual to an increased likelihood of physical disability, falls/fractures and mortality. Whilst sarcopenia is multifaceted and has no sole cause, reduced responses to environmental stimuli (namely nutrition (i.e. protein feeding) and exercise) termed "anabolic resistance", appears to be a governing role in the progression of age-related muscle atrophy. The maintenance of muscle mass is regulated by the dynamic relationship between muscle protein synthesis (MPS) and muscle protein breakdown (MPB) with anabolic resistance, therefore, centering upon the blunting of increases in MPS and/or suppression of MPB.

Aged muscle has consistently shown depressed MPS rates following feeding and also exercise when compared to young muscle. Additionally, older individuals need to consume a greater amount of protein compared to younger individuals to drive an MPS increase above baseline levels. This can often prove difficult due to older adults exhibiting increased satiety, likely contributing to the inadequate daily consumption of protein in such populations. Fortifying protein with leucine may, therefore, provide a nutraceutical avenue for combating anabolic resistance in ageing muscle. Leucine, both an essential amino acid (EAA) and branched chain amino acid (BCAA), is the key AA for stimulating MPS via activation of mechanistic target of rapamycin complex 1 (mTORC1), meaning protein rich in leucine may be advantageous to trigger MPS. Recent work has shown that a submaximal protein (10 g) drink enriched with leucine (4.5 g), compared to the non-essential amino acid (NEAA)- alanine (4.5 g), elevated MPS in older individuals, with anabolic signalling also being robustly triggered when administering ~6g BCAAs contain ~2.6 g leucine in older adults. However, research has also shown that in the absence of a full AA profile, leucine alone failed to stimulate MPS in postmenopausal women. It, therefore, remains inconclusive whether standalone or adjuvant supplementation of leucine is most effective to sufficiently stimulate MPS across aged populations and it remains to be investigated whether submaximal doses of complete protein enriched with leucine may lead to enhanced muscle anabolism in older adults.

In this study, we aim to assess the impact of dietary supplementation with a "super-whey" (SW) protein (with ~40% enhanced leucine and ~20% enhanced EAAs) vs. isonitrogenous whey protein (WP) on muscle protein synthesis (MPS). We will examine these effects both in the rested state, as well as the 24 hour post-exercise period under tightly controlled activity and feeding conditions.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* A BMI <18 or >35 kg/m2
* Active cardiovascular, cerebrovascular or respiratory disease: e.g. uncontrolled hypertension (BP > 160/100), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt, recent cardiac event, COPD, pulmonary hypertension or recent (6 mo) stroke
* Any metabolic disease
* Clotting dysfunction
* A history of, or current neurological or musculoskeletal conditions (e.g. epilepsy)
* Lactose intolerance
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Male participants are eligible for this study.
Enrollment: 30 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Muscle Protein Synthesis | From enrollment there is a three day lead in to the study with a controlled diet and limited physical activity, followed by two and a half days of study visits.
  We measure myofibrillar fractional synthesis rates (FSR) based on the incorporation of deuterated hydrogen from heavy water (D2O) in the muscle. Participants will consume the heavy water the day before the onset of the study, and then muscle biopsies will be taken at various points over the next three days for rested and post-exercise muscle protein synthesis measures.

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Atherton, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital Medical School, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No